CLINICAL TRIAL: NCT06235814
Title: Molecular Analysis for Precision Surgery in Thyroid Cancer (MAPS) Trial
Brief Title: Molecular Analysis for Precision Surgery in Thyroid Cancer Trial
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Masha Livhits, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#23-001404
Record Dates: First submitted 2024-01-18; First posted 2024-02-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Papillary Thyroid Cancer
Keywords: Radioactive Iodine; Fine Needle Aspiration; Parathyroid Hormone; Thyroid Stimulating Hormone; Thyroglobulin
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid Lobectomy (Active Comparator): Randomization Protocol
  Patients with intermediate molecular-risk thyroid nodules will be randomized to thyroid lobectomy or total thyroidectomy. We will perform a 1:1 randomization in a consecutive manner. Patients will be informed of what operation they will receive and providers will also be aware what operation was performed as it dictates care moving forward. Details of operative management will be discussed further.
  Peri-operative Protocol
  Thyroid Lobectomy Patients undergoing thyroid lobectomy will have the thyroid lobe containing the cancer removed in the standard surgical technique. These operations will be performed at either the UCLA Health Westwood Ambulatory Surgery Center, UCLA Ronald Reagan Medical Center, or UCLA Santa Monica Medical Center. Patients will undergo our usual postoperative care.
  Interventions: Procedure: Molecular Analysis for Thyroid Resection
- Total Thyroidectomy (Active Comparator): Randomization Protocol
  Patients with intermediate molecular-risk thyroid nodules will be randomized to thyroid lobectomy or total thyroidectomy. We will perform a 1:1 randomization in a consecutive manner. Patients will be informed of what operation they will receive and providers will also be aware what operation was performed as it dictates care moving forward. Details of operative management will be discussed further.
  Total Thyroidectomy and Completion Thyroidectomy
  Patients undergoing total thyroidectomy will have their whole thyroid gland removed in the standard surgical technique. Patients undergoing a completion thyroidectomy will have their remaining thyroid lobe removed. These operations will be performed at UCLA Ronald Reagan Medical Center or UCLA Santa Monica Medical Center. Patients will undergo our usual postoperative care.
  Interventions: Procedure: Molecular Analysis for Thyroid Resection

INTERVENTIONS:
Procedure: Molecular Analysis for Thyroid Resection — Protocol for Operative Management based on Molecular Risk Classifier
  Patients will have a televisit (i.e. video-visit) with us in 2 weeks once the ThyroSeq molecular analysis results. In that visit, we will discuss the operation the patient will receive, including the risks and benefits of the operation. Operative management will be dictated by the molecular results listed below:
  * Low molecular-risk: thyroid lobectomy
  * High molecular-risk: total thyroidectomy
  * Intermediate molecular-risk: randomization to thyroid lobectomy or total thyroidectomy
  Of note, the respective operations for the low and high molecular-risk groups are standard of care.

SUMMARY:
Ideal surgical extent for differentiated thyroid cancer remains unclear. Routine use of molecular analysis in biopsy-proven thyroid cancer could provide important prognostic information to help guide extent of surgery - thyroid lobectomy versus total thyroidectomy. This is a pilot feasibility study for the use of routine molecular analysis in Bethesda V and VI thyroid cancers, with randomization of the intermediate-molecular risk subgroup to thyroid lobectomy and total thyroidectomy. The investigators hypothesize that patients will 1) agree to preoperative molecular analysis, and 2) 50% of intermediate-risk patients will agree to and follow through with randomization. This will be a pilot study for a future randomized controlled trial (RTC) to compare between the two surgical approaches in intermediate-molecular risk thyroid cancer.

DETAILED DESCRIPTION:
Significance

Incidence of thyroid cancer has substantially increased in the past decade. Papillary thyroid cancers (PTC), typically follow a very indolent course. Although approximately 45,000 patients are diagnosed with thyroid cancer each year, only 2,000 patients die from it with a 5-year survival of over 98%. Thus, there has been a movement to de-escalate care to reduce unnecessary surgical morbidity, and current guidelines recommend consideration of thyroid lobectomy over total thyroidectomy when appropriate. At this time, it is unclear when thyroid lobectomy would be more beneficial than total thyroidectomy. A systematic review of guidelines and expert consensuses from 2009 to 2019 for PTC 1-4 cm in size found that 11 studies recommended total thyroidectomy, 5 recommended thyroid lobectomy, and 3 recommended either depending on patient-centered decision making. Thus, there is an unmet clinical need for improved preoperative risk stratification to determine ideal surgical treatment of thyroid cancer.

Currently, molecular testing is used to determine the risk of malignancy in indeterminate thyroid biopsies. However, these tests have not been used for prognostic purposes in biopsy-proven thyroid cancer. Recent studies have demonstrated that molecular profiling of thyroid cancer is predictive of recurrent disease. Certain high-risk mutations such as TP53, BRAF, and TERT are associated with increased risk of recurrence and fatal disease. Therefore, molecular testing can offer valuable prognostic information to guide treatment.

The investigators propose a feasibility study of a future multicenter study to assess routine use of preoperative molecular testing for risk stratification. The investigators believe that future studies stemming from this proposal will show that for patients with intermediate molecular risk PTC, thyroid lobectomy will have equivalent cancer outcomes to total thyroidectomy. If true, this will reduce the surgical risk and improve quality of life of the tens of thousands of thyroid cancer patients, without compromising cancer outcomes. Ultimately, the investigators hope to reduce overtreatment and morbidity in the treatment of this indolent disease.

Innovation

Routine use of molecular analysis in all thyroid cancer cases. The investigators propose to perform Thyroseq molecular testing on all patients who present with biopsy proven thyroid cancer. Routine molecular testing on a consecutive, prospective cohort will reveal the distribution of gene mutations and rearrangements in a diverse thyroid cancer population. Thyroseq, a DNA-RNA sequencing test of 112 thyroid cancer-associated genes, can provide state of the art data to help guide appropriate treatment for these patients.

Risk stratification for recurrence based on molecular analysis. Using Thyroseq's pre-determined risk of recurrence based on types of mutations present, the patients will be stratified as low-, intermediate-, or high-molecular risk. Several studies have demonstrated that certain combination of mutations, such as TERT/TP53, confer a significantly higher risk of mortality and recurrence, whereas BRAF mutations have been debated about their prognostic significance. Thus, the database generated from this risk stratification process will provide vital data regarding pathologic outcomes associated with these mutations.

Randomization for intermediate-risk PTC patients to thyroid lobectomy versus total thyroidectomy. Current ATA guidelines allow thyroid lobectomy or total thyroidectomy for PTCs 1-4 cm in size. The investigators are proposing one of the first studies to randomize patients with intermediate risk disease. This is the most robust method to determine whether outcomes are similar between thyroid lobectomy and total thyroidectomy. Currently, no randomized trial data exists regarding this topic.

Background

Diagnosis of thyroid cancer. Patients with thyroid nodules that look concerning on ultrasound undergo fine needle aspiration biopsy. These are then classified into the Bethesda Category based on risk of malignancy. Bethesda I is non-diagnostic and repeat biopsy is required, and Bethesda II is benign. Bethesda III and IV are indeterminate nodules. With the new advances in molecular genetics, current guidelines endorse utilization of next generation sequencing for these nodules to further delineate the risk of malignancy. Bethesda V nodules have a high risk for malignancy, and Bethesda VI is diagnostic of a malignancy, so those patients require operative resection. Genetic analysis is not routinely performed for these nodules. This study will focus on patients with these Bethesda V and VI nodules.

Surgical treatment of PTC. PTC is the predominant pathologic type of thyroid cancer, accounting for 80-90% of all cases. Patients with diagnosed thyroid cancer should undergo ultrasound of the neck to assess for sonographic evidence of extrathyroidal spread and lymph node metastasis.6 Patients with nodules larger than 4cm, gross extrathyroidal extension (clinical T4), or clinically apparent metastatic disease to lymph nodes (clinical N1) or distant sites (clinical M1) should undergo total thyroidectomy and gross removal of all primary tumor.6 For cancers < 1 cm and without clinical evidence of disease spread, ATA recommends performing a thyroid lobectomy to reduce morbidity. However, patients who fall in the middle with nodules between 1cm and 4cm without evidence of disease spread, guidelines recommend either thyroid lobectomy or total thyroidectomy based upon disease features and patient preference.

Postoperative radioactive iodine for high-risk disease on pathology. Patients who ultimately end up with high-risk disease on pathology (extrathyroidal extension, numerous lymph node involvement, high-risk histologic features, etc.) undergo radioactive iodine (RAI) therapy. In order to receive RAI, patients must have a total thyroidectomy. Those who initially had thyroid lobectomy and pathology returns with high-risk disease undergo a completion thyroidectomy - removal of the remaining thyroid gland - prior to starting RAI. After completion of all treatment, patients can be surveilled with routine ultrasound and thyroglobulin levels.

Thyroseq molecular analysis. Molecular analysis models were trained with machine learning algorithm on both pathologies that were confirmed to be benign (Bethesda II) and malignant (Bethesda V and VI) to analyze which genes and mutations are associated with malignancy.8 Thyroseq is a DNA- and RNA-based next generation sequencing model of 112 genes.4 It reports the analysis in six different categories that range from negative to presence of high-risk mutation (Figure 1). Based on Thyroseq's risk stratification, nodules with certain combinations of TERT/TP53 with BRAF mutations are considered high risk for recurrence,3 and total thyroidectomy is recommended. Conversely, RAS-like mutations are associated with non-invasive follicular thyroid neoplasm with papillary-like nuclear features (NIFTP), or a very low-risk variant of papillary thyroid cancer.9 Thus, a thyroid lobectomy is recommended for these low-risk cases. However, there exists a gray area in the appropriate management of Hurthle cell-type mutation and BRAF-type mutation, where thyroid lobectomy or total thyroidectomy are both considered adequate treatments.

Aim 1. Determine feasibility of a future multi-center trial of routine preoperative molecular testing for papillary thyroid cancers to guide extent of therapy. The investigators will pilot a single-center trial performing preoperative molecular testing on all biopsy confirmed thyroid cancers. Goal is to assess the feasibility of a future multi-center trial to determine prognostic value of preoperative molecular analysis.

Study setting and population. Patients seeking initial consultation at UCLA for newly diagnosed thyroid cancer (Bethesda V and VI nodules) with localized disease will be recruited for the study. The UCLA Endocrine Center is a high-volume tertiary referral center for patients with thyroid cancer, performing 300 thyroid operations annually. Of these patients, approximately 200 patients per year have localized disease eligible for this study. Inclusion criteria: patients aged 18 or older, English-speaking, with a new diagnosis of thyroid cancer. Exclusion criteria: patients with extra-thyroidal spread or with cancers >4cm in size.

Data collection. Patients enrolled in the study will have their thyroid nodule biopsy samples sent for Thyroseq analysis. Based on the mutations reported by Thyroseq (Figure 1), patients will be stratified as low-, intermediate-, or high-risk. Intermediate-risk patients will further be randomized to thyroid lobectomy or total thyroidectomy, explained in Aim 2. Patient outcomes will be tracked, which will be further delineated in Aim 3.

Feasibility study. For feasibility studies of randomized control trials, a sample size of 24 to 50 patients is recommended.10 Investigators anticipate that an obstacle to study completion will be poor adherence rates to the study, particularly randomization of surgical treatment in the intermediate-risk group. If investigators enroll 100 patients with 50 patients randomized to the invention arm, investigators predict a 75% completion rate of study assessments within a 95% confidence interval of +/- 12%. Thus, the investigators' target enrollment will be 120 patients to allow up to a 20% dropout rate, with 50 randomized to the intervention arm. The main endpoints of the feasibility measures will include: 1) number of patients screened compared to patients enrolled, 2) rate of study completion, and 3) dropout rate.

Aim 2. Determine the percent of eligible patients that undergo randomization to thyroid lobectomy versus total thyroidectomy and complete assigned treatment. Patients with intermediate-risk molecular analysis results will be further randomized to the above intervention, to assess ideal extent of operative intervention in this population.

Treatment characteristics. Patients will receive the usual counseling, preoperative, and postoperative care for the respective operations. Those who undergo total thyroidectomy will have weight-based thyroid hormone replacement prescribed. All patients will be followed by endocrine surgery and endocrinology for thyroid function management and cancer surveillance.

Outcomes of interest. Outcomes of interest include proportion of patients who 1) agree to randomization compared to those who enrolled in the study, and 2) complete the treatment as assigned. As mentioned above, investigators predict that 50% of enrolled patients will agree to randomization, with a dropout rate of 20%.

Aim 3. Determine whether preoperative molecular testing predicts postoperative clinicopathologic findings. Patients enrolled in the study will have their clinical and pathologic outcomes tracked in our database to assess the effectiveness of molecular risk stratification in thyroid cancer.

Database creation. All postoperative data will be obtained with chart review. Pathologic outcomes of interest include TNM staging, evidence of micro- and macroscopic extrathyroidal spread, lymph node involvement, and high-risk pathologic features. Clinical outcomes include rate of conversion to completion thyroidectomy in those who initially undergo lobectomy, rates of postoperative RAI therapy, and evidence of recurrence on imaging or laboratory values.

Effectiveness of molecular risk stratification. Ultimately, investigators will use multivariable logistic regression analysis to assess of the low-, intermediate-, and high-risk stratification correlate to final pathology outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older at the time of enrollment
* English-speaking
* Bethesda V or VI thyroid nodule that are 1-4cm in size
* Bethesda III or IV nodules who underwent previously underwent Thyroseq molecular analysis that returned with intermediate molecular risk disease

Exclusion Criteria:

* Prior thyroid operation
* Extrathyroidal extension or lymph node metastases seen on ultrasound
* Distant metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of eligible patients who enroll | 2 years
  Aim 1. Determine feasibility of a future multi-center trial of routine preoperative molecular testing for papillary thyroid cancers to guide extent of therapy. Patients with a new diagnosis of papillary thyroid cancer will undergo routine molecular testing with Thyroseq genomic classifier. Inclusion criteria include age over 18 years and cytology consistent with papillary thyroid cancer. We will exclude patients with hard indications for total thyroidectomy on ultrasound imaging (nodal or distant metastases, extrathyroidal extension). Patients' thyroid cancer molecular profile will be classified as low-, intermediate-, or high-risk based on previous published data.4 Endpoints are related to feasibility of a future trial. Main endpoint will be enrollment rate among eligible patients.

SECONDARY OUTCOMES:
Rate of patients who complete treatment as assigned | 2 years
  Aim 2. Determine the percent of eligible patients that undergo randomization to thyroid lobectomy versus total thyroidectomy and complete assigned treatment. There is equipoise between thyroid lobectomy and total thyroidectomy for intermediate risk molecular profile thyroid cancers. Thus, we will randomize those patients to thyroid lobectomy or total thyroidectomy. However, many patients may object to randomization or may not be willing to undergo treatment as randomized. Thus, we will assess percentage of patients who 1) agree to randomization, and 2) complete treatment as assigned. For patients who decline randomization or do not complete treatment, we will perform semi-structured exit interviews.
Rate of escalation of care from initially assigned treatment | 2 years
  Aim 3. Determine whether preoperative molecular testing predicts postoperative clinicopathologic findings. We will create a registry tracking the final surgical pathology and clinical results. Postoperative pathologic findings following thyroid surgery will be obtained using chart-review. We will determine whether certain mutations or intermediate or high risk molecular profiles predict the presence of pathologic features that benefit from radioiodine treatment. Additionally, we will track postoperative cancer surveillance outcomes, including recurrence seen on imaging and laboratory values.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT06235814/Prot_SAP_001.pdf